CLINICAL TRIAL: NCT01818375
Title: Goal-directed Fluid Therapy and Postoperative Ileus After Elective Laparoscopic Colorectal Surgery Using an Enhanced Recovery Program: a Randomized Controlled Trial
Brief Title: Goal Directed Fluid Therapy and Postoperative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriele Baldini, MD, MSc, Assistant Professor (Other)
Responsible Party: Sponsor-Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, MD, MSc, Anesthesiologist, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 12-277-SDR
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal Directed Fluid Therapy (GDFT) (Experimental): During surgery, patients in the Goal Directed Fluid Therapy (GDFT) will receive:
  1. maintenance infusion of intravenous infusion of ringer lactate at a rate of 1.5 ml/Kg/hr to compensate insensible blood loss and fluid shift during surgery as recommended by perioperative fluid management guidelines for patients undergoing surgery with an enhanced recovery program and receiving a GDFT approach;
  2. intraoperative intravenous boluses of colloids (6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride-Voluven) guided by an algorithm based on Esophageal Doppler (ED) estimation of the stroke volume (SV) provided by the manufacture, and also used in other clinical trials.
  Interventions: Procedure: Goal Directed Fluid Therapy (GDFT)-Esophageal doppler guided
- Standard Fluid Therapy (Active Comparator): During surgery, patients will receive a maintenance infusion of intravenous infusion of ringer lactate as recommended by international guidelines and anesthesia text-books (Standard Fluid Therapy). In the Standard Fluid Therapy arm, the Esophageal Doppler (ED) monitor will be turned away from the anesthesia care provider, and the screen will be covered with an opaque card. The ED variables will be collected by an independent research personnel. Hemodynamic variables triggering extra fluid administration (Ringer Lactate or Voluven) will be decided based on the clinical judgment of the anesthetist in charge and will include: urinary output less than 0.5/ml/kg/hr, an increase in heart rate more than 20% above baseline or more than 110 beats/min, a decrease in mean systolic blood pressure less than 20% below baseline or less than 90 mmHg and intraoperative blood loss. Boluses of 200 ml of intravenous fluid will be administered until the above targets will be restored
  Interventions: Other: Standard fluid therapy

INTERVENTIONS:
Procedure: Goal Directed Fluid Therapy (GDFT)-Esophageal doppler guided
  Other Names: Esophageal doppler-Deltex Medical
  Arms: Goal Directed Fluid Therapy (GDFT)
Other: Standard fluid therapy
  Other Names: Intravenous infusion as recommended by international guidelines and anesthesia text-books
  Arms: Standard Fluid Therapy

SUMMARY:
Despite Goal Directed Fluid Therapy (GDFT) has shown a reduction of hospitalization and overall complications in patients undergoing abdominal surgery, there is a need to address the effect of implementing GDFT on the incidence of specific surgical complications and in a context of en enhanced recovery program (ERP). Specifically, studies investigating the impact of GDFT on primary postoperative ileus (POI) in patients undergoing laparoscopic colorectal surgery and using an ERP are missing.

It is hypothesized that the incidence of primary POI will be reduced in patients receiving intraoperative GDFT compared to patients receiving Standard Fluid Therapy (SFT) after elective laparoscopic colorectal surgeries with an ERP program.

DETAILED DESCRIPTION:
Randomized Controlled Trial. Study population: elective laparoscopic colorectal resections with an Enhanced Recovery Program (ERP) Sample size: 128 patients (140 accounting for drops out)

Two arms:

GDFT: patients will receive GDFT esophageal doppler guided; SFT: patients will receive SFT based on standard anesthesia formula and international guidelines to calculate fluid requirements.

Study Hypothesis: the incidence of primary POI will be reduced in patients receiving intraoperative GDFT compared to patients receiving SFT after elective laparoscopic colorectal surgeries with an ERP program.

ERP: all patients will receive the same perioperative care according to the Enhanced Recovery After Surgery ERAS® program guidelines. Intravenous fluid will be stopped the first day after surgery. Patients will be allowed to have clear fluids the same day of surgery and diet, as tolerated, the first day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective laparoscopic colorectal resection with an Enhanced Recovery Program

Exclusion Criteria:

1. Age <18 yr
2. Emergency surgery
3. Patients who do not understand, read or communicate in either French or English
4. Patients who had undergone esophageal or gastric surgery
5. Esophageal pathology (esophageal varices or cancer)
6. Patients with coarctation of the aorta or aortic stenosis
7. Chronic atrial fibrillation

7. Preoperative bowel obstruction 8. Coagulopathies 9. Chronic use of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Primary postoperative ileus (POI) | participants will be followed for the duration of hospital stay, an expected average of 3 days
  Patients will be considered having primary POI if at least one symptom, for each of the following criteria, will be reported:
  i. vomiting (+/- nausea) OR abdominal distension AND ii. Absence of passing gas/stool OR not tolerating oral diet.

SECONDARY OUTCOMES:
Intraoperative hemodynamic measurements | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Systolic blood pressure; diastolic blood pressure; mean arterial blood pressure; heart rate; flow-time corrected (FTc); stroke distance (SD); Peak velocity (PV); stroke volume (SV); stroke index (SVI); cardiac output (CO); cardiac Index (CI)
Intraoperative and postoperative fluids and blood products required | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Vasoactive agents required | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Urinary output | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Intraoperative and postoperative urinary output | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Intraoperative and Postoperative opioid consumption | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Intraoperative opioid administration and postoperative opioid consumption
Postoperative nausea and vomiting (PONV) | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Time spent out of bed | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Postoperative complications (Clavien Classification) | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Patients' weight | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Quality of surgical recovery score | Participants will be followed for the duration of hospital stay, an expected average of 3 days
Readiness to be discharged | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  : according to the colorectal pathway, hospital discharge is planned on postoperative day 3. Patients will be discharged if afebrile, able to tolerate oral diet, pain is controlled (NRS < 4), and able to ambulate
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Challand C, Struthers R, Sneyd JR, Erasmus PD, Mellor N, Hosie KB, Minto G. Randomized controlled trial of intraoperative goal-directed fluid therapy in aerobically fit and unfit patients having major colorectal surgery. Br J Anaesth. 2012 Jan;108(1):53-62. doi: 10.1093/bja/aer273. Epub 2011 Aug 26. PMID 21873370
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Rahbari NN, Zimmermann JB, Schmidt T, Koch M, Weigand MA, Weitz J. Meta-analysis of standard, restrictive and supplemental fluid administration in colorectal surgery. Br J Surg. 2009 Apr;96(4):331-41. doi: 10.1002/bjs.6552. PMID 19283742
- [Background] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):801-16. doi: 10.1016/j.clnu.2012.08.012. Epub 2012 Sep 26. PMID 23062720
- See also: Related Info — http://www.deltexmedical.com/